CLINICAL TRIAL: NCT00666172
Title: Effects of Worksite Wellness Interventions on Vascular Function, Insulin Sensitivity and High-Density Lipoprotein in Overweight or Obese Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 080108; 08-H-0108
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-08-18

CONDITIONS: Atherosclerosis; Diabetes Mellitus; Obesity; Dyslipidemia; Hypertension
Keywords: Women's Health; Obesity; Metabolic Syndrome; Arterial Function; Lipoproteins; Overweight
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus; Obesity; Dyslipidemias; Hypertension; Metabolic Syndrome; Overweight | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise
Behavioral: Weight Loss

SUMMARY:
Employees in developed societies are becoming increasingly sedentary at work and at home due to technological advances. Physical inactivity coupled with excess intake of calorie-rich foods are responsible for the epidemic of obesity. In population cohorts, physical inactivity and obesity increase the risk of cardiovascular disease and death. Because of the impact on productivity and health care costs, many businesses and other organizations have initiated "wellness" programs, often with facilities at the work site to encourage exercise. Although these programs have often resulted in improved fitness for participants, weight loss has been more difficult to achieve. In this regard, in our initial study of NIH employees participating in NHLBI's Keep the Beat program--two-thirds of whom were overweight or obese--we found improved exercise fitness after 3 months of participation, with exercise averaging 20 minutes each work day, but no significant weight loss. Associated with greater fitness in our participants was improvement in endothelial function, an important biomarker of cardiovascular risk. Because level of fitness is a strong predictor of cardiovascular (and total) mortality in population studies, some investigators and thought leaders have proposed that it is acceptable to be "fat and fit." We found in our study, however, that exercise alone has little effect on insulin sensitivity and other biomarkers of risk, including C-reactive protein, which could limit further improvement in endothelial function and even greater risk reduction. We propose to test in this protocol whether weight loss through supervised nutritional counseling and daily exercise at worksite facilities confers health benefits beyond those achieved with improved fitness alone, such as improvement in endothelial function, arterial compliance, insulin sensitivity, markers of inflammation in blood and high-density lipoprotein (HDL) structure and function. Because obesity in a sedentary workforce environment is especially prevalent among women, with additional contribution of menopause to obesity, our study will be restricted to overweight and obese women to allow appropriate analysis in a cohort of manageable size for our testing resources. The primary endpoint will be differential improvement in endothelial function, as determined by brachial artery reactivity to shear stress, from baseline to 6 months in participants randomized to exercise coupled with weight-loss intervention versus subjects randomized to exercise alone. Secondary analyses will include comparisons of adiposity, arterial stiffness, insulin sensitivity, HDL subparticles and function, and markers of inflammation and adipokines in blood, with exploratory analyses of minorities and age/hormonal interactions. Demonstration of improved vascular function and other biomarkers of cardiovascular risk with improved fitness combined with weight loss may serve as an incentive for greater participation in organization-initiated wellness programs with emphasis both on exercise and on personalized nutritional counseling.

DETAILED DESCRIPTION:
Employees in developed societies are becoming increasingly sedentary at work and at home due to technological advances. Physical inactivity coupled with excess intake of calorie-rich foods are responsible for the epidemic of obesity. In population cohorts, physical inactivity and obesity increase the risk of cardiovascular disease and death. Because of the impact on productivity and health care costs, many businesses and other organizations have initiated "wellness" programs, often with facilities at the work site to encourage exercise. Although these programs have often resulted in improved fitness for participants, weight loss has been more difficult to achieve. In this regard, in our initial study of NIH employees participating in NHLBI's Keep the Beat program--two-thirds of whom were overweight or obese--we found improved exercise fitness after 3 months of participation, with exercise averaging 20 minutes each work day, but no significant weight loss. Associated with greater fitness in our participants was improvement in endothelial function, an important biomarker of cardiovascular risk. Because level of fitness is a strong predictor of cardiovascular (and total) mortality in population studies, some investigators and thought leaders have proposed that it is acceptable to be "fat and fit." We found in our study, however, that exercise alone has little effect on insulin sensitivity and other biomarkers of risk, including C-reactive protein, which could limit further improvement in endothelial function and even greater risk reduction. We propose to test in this protocol whether weight loss through supervised nutritional counseling and daily exercise at worksite facilities confers health benefits beyond those achieved with improved fitness alone, such as improvement in endothelial function, arterial compliance, insulin sensitivity, markers of inflammation in blood and high-density lipoprotein (HDL) structure and function. Because obesity in a sedentary workforce environment is especially prevalent among women, with additional contribution of menopause to obesity, our study will be restricted to overweight and obese women to allow appropriate analysis in a cohort of manageable size for our testing resources. The primary endpoint will be differential improvement in endothelial function, as determined by brachial artery reactivity to shear stress, from baseline to 6 months in participants randomized to exercise coupled with weight-loss intervention versus subjects randomized to exercise alone. Secondary analyses will include comparisons of adiposity, arterial stiffness, insulin sensitivity, HDL subparticles and function, and markers of inflammation and adipokines in blood, with exploratory analyses of minorities and age/hormonal interactions. Demonstration of improved vascular function and other biomarkers of cardiovascular risk with improved fitness combined with weight loss may serve as an incentive for greater participation in organization-initiated wellness programs with emphasis both on exercise and on personalized nutritional counseling.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Female employees of NIH who are not currently participating or greater than 3 months from participation in the Keep the Beat program or other structured exercise or weight-loss program (e.g., Weight Watchers, NutriSystems, personalized nutritional counseling or fitness trainers), and have not undergone weight loss (bariatric) surgery. Self-directed exercise (walks around the block, climbing stairs) is acceptable for inclusion, with subjects encouraged to continue such activity, in addition to worksite exercise, throughout the program.
  2. Body-mass index greater than or equal to 25 kg/m(2).
  3. Subject understands protocol and provides written, informed consent in addition to willingness to comply with specified follow-up evaluations.

EXCLUSION CRITERIA:

1. Medical condition, including recent unintentional weight loss, that might prohibit safe participation in the Keep the Beat program.
2. Fluctuation in weight greater than 5 percent over previous 3 months by self report.
3. Fasting blood glucose greater than or equal to 126 mg/dL in absence of prior diagnosis of diabetes mellitus.
4. Weight greater than 200 kg (exceeds capacity of DXA scanner).
5. Heart disease as indicated by history of myocardial infarction, documented disease on coronary angiography, coronary artery stent placement, congestive heart failure, significant structural heart disease (e.g. hypertrophic or dilated cardiomyopathy, valvular heart disease).
6. Hyper- or hypothyroid by routine lab screening.
7. Physically unable to perform the Keep the Beat program due to neurologic or orthopedic conditions.
8. Pregnant women due to large hormonal changes in pregnancy that affect study variables and potential pregnancy-related restrictions on exercise.
9. Participation in another study protocol which includes blood draws or interventions.
10. Use of medications that might interfere with, or promote, weight loss.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2008-04-08; Primary Completion 2012-11-01 (Actual); Study Completion 2012-11-01 (Actual)

PRIMARY OUTCOMES:
Measure endothelial function determined by brachial artery reactivity to stress, at baseline/following 6m program participation comparison of change between subj randomized to exercise with weight-loss intervention vs. those randomized to exerci...

CONTACTS AND LOCATIONS:
Overall Officials: Richard O Cannon, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ludmer PL, Selwyn AP, Shook TL, Wayne RR, Mudge GH, Alexander RW, Ganz P. Paradoxical vasoconstriction induced by acetylcholine in atherosclerotic coronary arteries. N Engl J Med. 1986 Oct 23;315(17):1046-51. doi: 10.1056/NEJM198610233151702. PMID 3093861
- [Background] Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR Jr, Lerman A. Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. Circulation. 2000 Mar 7;101(9):948-54. doi: 10.1161/01.cir.101.9.948. PMID 10704159
- [Background] Schachinger V, Britten MB, Zeiher AM. Prognostic impact of coronary vasodilator dysfunction on adverse long-term outcome of coronary heart disease. Circulation. 2000 Apr 25;101(16):1899-906. doi: 10.1161/01.cir.101.16.1899. PMID 10779454